CLINICAL TRIAL: NCT00071942
Title: A Phase I Trial of An Admixture of Recombinant Vaccinia Virus That Express DF3/MUC1 and rV-TRICOM (B7.ICAM-1, and LFA-3) in Patients With Metastatic Adenocarcinoma of The Breast
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03131; NCI-2012-03131 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); DFCI-02310; NCI-5747; 02-310 (Other: Dana-Farber Cancer Institute); 5747 (Other: CTEP); U01CA062490 (NIH); NCT00077571 (obsolete NCT alias)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — rV-Tricom

ARMS (1):
- Treatment (vaccine therapy) (Experimental): Patients receive vaccination comprising recombinant vaccinia-MUC-1 and recombinant vaccinia-TRICOM vaccine intradermally on days 1 and 29 (for a total of 2 doses) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: recombinant vaccinia-MUC1 vaccine; Biological: recombinant vaccinia-TRICOM vaccine; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment

INTERVENTIONS:
Biological: recombinant vaccinia-MUC1 vaccine — Given intradermally
  Other Names: recombinant vaccinia-MUC-1 vaccine; rV-MUC-1; vaccinia-MUC-1 vaccine
Biological: recombinant vaccinia-TRICOM vaccine — Given intradermally
  Other Names: rV-TRICOM; Vaccinia-TRICOM
Other: laboratory biomarker analysis — Correlative studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
Vaccines may make the body build an immune response to kill tumor cells. This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the toxicity associated with repeated vaccination with an admixture of recombinant vaccinia viruses (rV-MUC-1 and rV-TRICOM).

II. To determine the maximum tolerated dose (MTD) of rV-MUC-1 and rV-TRICOM vaccine admixture.

III. To evaluate the toxicity of adding GM-CSF to the admixture of the rV-MUC-1 and rV-TRICOM.

SECONDARY OBJECTIVES:

I. To assess host immune reactivity following rV-MUC-1 and rV-TRICOM with and without GM-CSF administration.

II. To determine whether vaccination with rV-MUC-1 and rV-TRICOM with and without GM-CSF is associated with antitumor activity.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive vaccination comprising recombinant vaccinia-MUC-1 and recombinant vaccinia-TRICOM vaccine intradermally on days 1 and 29 (for a total of 2 doses) in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of recombinant vaccinia-MUC-1 and recombinant vaccinia-TRICOM vaccine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 10 patients (including 5 HLA-A2-positive patients) receive vaccination as above at the MTD and sargramostim (GM-CSF) subcutaneously on days 1-4 and 29-32.

Patients are followed at 4 weeks, monthly until disease progression, and then annually for up to 15 years.

PROJECTED ACCRUAL: A total of 11-22 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologically confirmed diagnosis of metastatic carcinoma of the breast; measurable disease is not required; subjects who are NED are eligible; subjects must have had at least one prior regimen of chemotherapy, immunotherapy, or hormonal therapy prior to entering this study; subjects may have received any number of prior therapies for metastatic disease
* Subjects must have an ECOG performance status of 0-1
* WBC > 2000/mm^3
* Platelet count > 100,000/mm^3
* Serum creatinine =< 2.0 mg/dl
* Serum bilirubin =< 1.5 mg/dl
* SGPT < 3 times the upper limit of normal
* >= 4 weeks since chemotherapy (>= 6 weeks for nitrosoureas or mitomycin C), hormonal therapy or radiation therapy; subjects must have recovered from all acute toxicity associated with the prior regimen; subjects receiving concurrent hormonal treatment or local radiation are not eligible
* Subjects must be HLA typed if not already previously done (5/10 subjects at the MTD dose level must be HLA A2 positive)
* Subjects must not have clinical evidence of altered immune responsiveness or autoimmune syndromes (scleroderma, systemic lupus erythematosus, etc.); subjects must be HIV antibody negative; this treatment may be associated with increased adverse effects for individuals with immune deficiencies, and HIV-associated symptoms preclude accurate assessment of toxicity
* Subjects must not have undergone splenectomy
* The recombinant vaccinia vaccine should not be administered if the following apply to either recipients or, for at least three weeks after vaccination, their close household contacts: persons with active or a history of extensive eczema or other eczematoid skin disorders; those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne or other open rashes or wounds) until condition resolves; pregnant or nursing women; children under 5 years of age; and immunodeficient or immunosuppressed persons (by disease or therapy), including HIV infection; close household contacts are those who share housing or have close physical contact; determination of the severity of these conditions will be made by the investigator or co-investigator
* Subjects must not have any other serious medical condition that in the opinion of the investigator is incompatible with the protocol; subjects with active infections requiring antibiotics are not eligible until the infection has cleared and the antibiotics have been stopped for at least 3 days
* Subjects must have had prior vaccinia (smallpox) exposure, determined by subject history, medical documentation, or scar characteristic of vaccinia exposure; there must be no history of allergy or untoward reaction to prior vaccinia (smallpox) vaccination
* Tumor tissue positive for staining with MAbs DF3 and/or DF3-P or elevated serum CA15-3 (also known as CA27-29); note: this can be done on stored slides, but subject will be responsible for costs if not covered by insurance
* Subjects must not have a history of seizures, encephalitis or multiple sclerosis
* Subjects must not be allergic to eggs
* Women of child-bearing potential must agree to use highly effective contraception or abstinence prior to study entry and for at least 4 weeks after the last vaccination; women who are breast-feeding are not eligible for this study; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Signed informed consent
* Participants who have been previously treated with vaccinia vectors or MUC1 such as those on protocol T98-0057 (DFPCC # 97-050) are not eligible for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2003-10; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose level preceding the dose in which 2 out of 6 patients experience dose limiting toxicity (DLT) assessed using National Cancer Institute (NCI) Common Toxicity Criteria version 2.0 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Eder, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States